CLINICAL TRIAL: NCT03417388
Title: Women's IschemiA TRial to Reduce Events In Non-ObstRuctive CAD
Acronym: WARRIOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201701142 -A; W81XWH-17-2-0030 (Other Grant/Funding Number: Department of Defense); OCR17268 (Other: UF OnCore); IRB201802734 (Other: UF IRB + VA); IRB201701434 (Other: UF IRB-01)
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Angiography; Coronary CT Angiogram; Ischemia; Non-obstructive CAD
MeSH Terms: conditions — Coronary Artery Disease; Ischemia | interventions — Atorvastatin; Rosuvastatin Calcium; Lisinopril; Losartan; Aspirin

STUDY DESIGN:
Intervention Model Description: This will be a PROBE design, that will evaluate an intensive statin/ACE-I (or ARB) plus ASA if tolerated, treatment strategy (IMT) vs. primary prevention risk factor therapy treatment strategy (UC) in symptomatic (chronic angina or equivalent) women with non-obstructive CAD.
Who Masked: Outcomes Assessor
Masking Description: The Clinical Events Committee (CEC) will be masked to all treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive Medical Treatment (IMT) (Experimental): The IMT-assigned women will receive high dose potent statin, and moderate dose of an ACE-I (lisinopril) or ARB (losartan). Aspirin will also be recommended to IMT women without contraindications or bleeding risk. This group will also receive Lifestyle Counseling (PACE Assessment), Quality of Life questionnaires, and the same visit schedule and "face-time" with site staff to reduce bias.
  Interventions: Drug: High dose potent statin; Drug: ACE-I (lisinopril) or ARB (losartan); Drug: Aspirin 81 enteric coated tablet daily; Behavioral: Lifestyle Counseling; Behavioral: Quality of Life Questionnaires
- Usual Care (UC) (Active Comparator): The UC-assigned women will maintain standard of care. This group will also receive Lifestyle Counseling (PACE Assessment), Quality of Life questionnaires, and the same visit schedule and "face-time" with site staff to reduce bias.
  Interventions: Behavioral: Quality of Life Questionnaires

INTERVENTIONS:
Drug: High dose potent statin — The IMT-assigned women will receive high-dose, potent statin (atorvastatin 40-80 mg/d or rosuvastatin 20-40mg) class of lipid-lowering medications.
  Other Names: atorvastatin or rosuvastatin
  Arms: Intensive Medical Treatment (IMT)
Drug: ACE-I (lisinopril) or ARB (losartan) — Angiotensin converting enzyme inhibitors (ACE inhibitors) and angiotensin receptor blockers (ARBs) are widely prescribed for primary hypertension.
  Other Names: ACE-I or ARB
  Arms: Intensive Medical Treatment (IMT)
Drug: Aspirin 81 enteric coated tablet daily — Will be recommended to IMT women without contraindications or bleeding risk.
  Other Names: Aspirin
  Arms: Intensive Medical Treatment (IMT)
Behavioral: Lifestyle Counseling — The PACE Lifestyle Assessment Intervention which is a program to assist with smoking cessation, weight loss, and exercise.
  Other Names: PACE Lifestyle Intervention
  Arms: Intensive Medical Treatment (IMT)
Behavioral: Quality of Life Questionnaires — Quality of Life Questionnaires will be obtained.
  Other Names: QOL

SUMMARY:
The Ischemia-IMT (Ischemia-Intensive Medical Treatment Reduces Events in Women with Non-Obstructive CAD), subtitle: Women's Ischemia Trial to Reduce Events in Non-Obstructive CAD (WARRIOR) trial is a multicenter, prospective, randomized, blinded outcome evaluation (PROBE design) evaluating intensive statin/ACE-I (or ARB)/aspirin treatment (IMT) vs. usual care (UC) in 4,422 symptomatic women patients with symptoms and/or signs of ischemia but no obstructive CAD. The hypothesis is that IMT will reduce major adverse coronary events (MACE) 20% vs. UC. The primary outcome is first occurrence of MACE as death, nonfatal MI, nonfatal stroke/transient ischemic attack (TIA) or hospitalization for heart failure or angina. Secondary outcomes include quality of life, time to "return to duty"/work, health resource consumption, angina, cardiovascular (CV) death and primary outcome components. Events will be adjudicated by an experienced Clinical Events Committee (CEC). Follow-up was planned to be 3-years using 50 sites: primarily VA and Active Duty Military Hospitals/Clinics and a National Patient-Centered Clinical Research Network (PCORnet) clinical data research network (CDRN)(OneFlorida Consortium). The number of sites were increased and follow up was modified to continue until the last patient enrolled was followed until trial follow up was completed. Recruitment was complete January 6, 2024.

This study is being conducted to determine whether intensive medication treatment to modify risk factors and vascular function in women patients with coronary arteries showing no flow limit obstruction but with cardiac symptoms (i.e., chest pain, shortness of breath) will reduce the patient's likelihood of dying, having a heart attack, stroke/TIA or being hospitalized for cardiac reasons. The results will provide evidence data necessary to inform future guidelines regarding how best to treat this growing population of patients, and ultimately improve the patient's cardiac health and quality of life and reduce health-care costs.

DETAILED DESCRIPTION:
WARRIOR trial is a multi-site, PROBE design, that will evaluate an intensive statin/ACE-I (or ARB)/aspirin treatment strategy (IMT) vs. primary prevention risk factor therapy treatment strategy (UC) in 4,422 symptomatic (chronic angina or equivalent) women with non-obstructive CAD (<50% diameter narrowing).

There will be ~80 US sites, including VA/ military and OneFlorida CDRN sites, with a proven record in prior trials. The investigators will use web-based, real-time data entry, and management University of Florida Data Management System (UFDMS) for site selection, screening, participant eligibility confirmation, enrollment, and randomization. Participants will be recruited from screened women with symptoms suspected to be ischemic with non-obstructive CAD by invasive coronary angiogram or CT angiogram. The high dose statin (atorvastatin or rosuvastatin) and ACE-I (lisinopril) [or ARB (losartan)] are generic commonly used medications previously demonstrated effective for improving angina, stress testing, myocardial perfusion and coronary microvascular flow reserve in small size trials in this population. Additionally, aspirin will also be recommended to IMT participants without contraindications or excess bleeding risk, however aspirin will not be provided by the study. Both the groups will also receive Lifestyle Counseling (PACE Assessment), and the same visit schedule and "face-time" with site staff to reduce bias. Events will be adjudicated by the Clinical Events Committee (CEC), according to objective criteria and masked to treatment assignment clues.

ELIGIBILITY:
Inclusion Criteria:

* Signs and symptoms of suspected ischemia prompting referral for further evaluation by cardiac catheterization or coronary angiogram or coronary CT angiogram within 5 years from consent
* Willing to provide written informed consent
* Non-obstructive CAD defined as 0 to 49% diameter reduction of a major epicardial vessel or a FFR>0.80

Exclusion Criteria:

* History of noncompliance (with medical therapy, protocol, or follow-up)
* History of non-ischemic dilated or hypertrophic cardiomyopathy
* Documented acute coronary syndrome(ACS) within previous 30 days
* Left ventricular ejection fraction (LVEF) <40%, New York Heart Association heart failure (NYHA HF) class III-IV, or hospitalization for Reduced ejection fraction (HFrEF) within 180 days
* Stroke within previous 180 days or intracranial hemorrhage at any time
* End-stage renal disease, on dialysis, or estimated glomerular filtration rate (eGFR) <30 ml/min.
* Severe valvular disease or likely to require surgery/Transcatheter aortic valve replacement (TVAR) within 3 years
* Life expectancy <3-yrs. due to non-cardiovascular comorbidity
* Enrolled in a competing clinical trial
* Prior intolerance to both an ACE-I and ARB
* If intolerant to a statin unless taking a PCSK9 as a statin replacement by their clinical provider
* Pregnancy (all pre-menopausal females must have negative urine pregnancy test if randomized to IMT before study drugs are prescribed. If they have not gone through menopause, had a hysterectomy, oophorectomy, or sterilization such as tubal ligation procedure)

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2476 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-09-14 (Actual)

PRIMARY OUTCOMES:
The primary outcome is MACE, defined as first occurrence of all-cause death, non-fatal MI, non-fatal stroke, or hospitalization for angina or HF. | Within 5 years
  All-cause death will be used 1) CV death is insensitive in this population with non-obstructive CAD since death is less likely attributed to CV causes when no obstructive CAD is present; 2) all-cause death is resistant to ascertainment bias in this unblinded trial. CV death will be defined broadly to include both definite CV death and possible CV death (all deaths except those with definite non-CV cause, e.g., cancer, witnessed trauma and homicide).
  The MI definition follows universal criteria for Types 1-5 MI events. Stroke/TIA definition is new onset neurological defect of central origin confirmed by brain imaging (CT or MRI) evidence of cerebral infarction or intracerebral hemorrhage.
  Hospitalization for angina- Any hospitalization for angina, plus unstable angina or ACS.
  Hospitalization for Heart Failure -required established objective criteria for heart failure.
  All MACE events are adjudicated by a blinded Clinical Endpoint Committee

SECONDARY OUTCOMES:
Components of MACE | Within 5 years
  The analysis will be repeated for the following combinations of MACE events (1) composite outcome of CV-death, non-fatal MI, or non-fatal stroke/TIA; (2) composite outcome CV-death, non-fatal MI, resuscitated cardiac arrest, or hospitalization for angina or heart failure; (3) all-cause mortality; (4) CV-death (5) total MI [fatal plus non-fatal]; (6) resuscitated cardiac arrest; (7) hospitalization for angina; (8) hospitalization for HF; (9) total stroke/TIA [fatal plus non- fatal]; (10) composite outcome of CV-death, non-fatal MI, stroke/TIA, resuscitated cardiac arrest, or hospitalization for angina or heart failure.
Composite hierarchical MACE endpoint | Within 5 years
  The comparison of randomized treatment strategies for composite hierarchical endpoint will be conducted using win statistics (WS), including the win ratio (WR), win odds (WO), will be computed to compare two groups based on hierarchical order of clinical importance as follows: 1) all cause death within 5 yrs, 2) stroke within 5 yrs, 3) MI within 5 yrs, 4) number of hospitalization within 5 yrs, 5) first hospitalization for heart failure or chest pain within 5 yrs, and 6) average of SAQ7 at 6 months and 1-year. The WR method compares each patient in the intervention group with every patient in the control group, and the magnitude of the effect is computed as the ratio of the total number of pairwise "wins" to "losses" considering the predefined hierarchy of the outcomes. Since the WR does not account for ties that the WO will also be computed. The benefit of the IMT arm is indicated by an estimate of WS/WO test statistic with their respective 95% confidence intervals greater than 1.
Seattle Angina Questionnaire (SAQ). | Study entry and every six months until end of follow up (up to 72 months)
  QoL comparisons will adhere to the ITT principle. We will examine changes over time from baseline and identify the major determinants of those changes using regression analysis. Questionnaires, such as the SAQ scores, at each time point will be analyzed using linear mixed models with correlation within subjects over time. In case the outcome residuals do not have a normal distribution, a transformation will be considered (e.g. log, Box-Cox). Interaction of group and time effects will be examined to assess for different time trends between groups.
EQ-5D-3L | Study entry and every six months until end of follow up (up to 72 months)
  Evaluated over time by group.
Duke Activity Status Inventory (DASI) | Study entry and every six months until end of follow up (up to 72 months)
  DASI as assessed over time by group.
Modified Morisky Medicine Scale Take your medication | Study entry and every six months until end of follow up (up to 72 months)
  Measure of medication compliance between groups over time.
PACE (Programs of All-Inclusive Care for the Elderly). | Study entry and every six months until end of follow up (up to 72 months)
  Assessment of healthy lifestyle intervention between groups over time.
PCL-5 (Screening for PTSD). | Study entry and every six months until end of follow up (up to 72 months)
  Screening for PTSD over time between groups
Health care utilization and cost effectiveness | Study entry and every six months until end of follow up (up to 72 months)
  Comparing health care resource utilization across time between groups.
GAD 7 | Study entry and every six months until end of follow up (up to 72 months)
  Assessment of general anxiety over time between groups
PHQ 8 | Study entry and every six months until end of follow up (up to 72 months)
  Assessment of depression over time between groups
MACE and Quality of Life outcomes will also be stratified by enrollment assessment of non-obstructive CAD using noninvasive CCTA vs invasive coronary angiography | Within 5 years
  MACE is first occurrence of all cause death, non fatal MI, non fatal stroke or TIA, hospitalization for heart failure, hospitalization for chest pain/angina. Quality of life is being assessed using Seattle Angina Questionnaire, SAQ7 and all of the SAQ domains, PTSD is being assessed using the PCL5, functional capacity is being assessed using the Duke Activity Status Index, EQ-5D-3L, Depression is being assessed using the PHQ-8 and anxiety using the GAD-7

OTHER OUTCOMES:
An analysis of MACE with repeated events considering the number of previous events as a time-dependent covariate will be performed | Within 5 years
  Using Andersen-Gill model with frailty to describe the repeated events: all-cause death, non-fatal MI, non-fatal stroke/TIA, or hospitalization for either angina or heart failure. Definitions of repeated events include 30 days between a documented MI and death as a standard definition for "Fatal MI" and >48hrs was a standard for exacerbation of ischemia (chest pain or ECG changes of ischemia) to call it a "new event" (e.g., either an MI, HF, or another exacerbation of ischemia).

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Pepine, MD, Principal Investigator — University of Florida
Locations (81):
- United States (80):
  - Cardiology Associates of Mobile, Inc., Mobile, Alabama
  - Dignity Health-Mercy Gilbert Medical Center, Gilbert, Arizona
  - Dignity Health-St. Joseph, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - University of Arkansas, Little Rock, Arkansas
  - Cedars-Sinai Heart Institute, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center, Torrance, California
  - Georgetown University, Washington D.C., District of Columbia
  - Clearwater Cardiovascular Consultants Clinical Research, Clearwater, Florida
  - South Palm Cardiovascular Research Institute, Delray Beach, Florida
  - Family Medicine at Eastside Community Practice, Gainesville, Florida
  - Family Medicine at Hampton Oaks Medical Plaza (Adults and Peds), Gainesville, Florida
  - Internal Medicine at Tower Hill, Gainesville, Florida
  - Family Medicine at Haile Plantation (Adults & Peds), Gainesville, Florida
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - Cardiovascular Clinic at UF Health UF, Gainesville, Florida
  - Internal Medicine at UF Health Medical Plaza, Gainesville, Florida
  - Spring Hill Cardiology, Gainesville, Florida
  - Family Medicine at 4th Ave, Gainesville, Florida
  - Family Medicine at Old Town (Adults and Peds), Gainesville, Florida
  - Baptist Health, Jacksonville, Florida
  - University of Florida, Jacksonville, Jacksonville, Florida
  - Naval Hospital Jacksonville, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - UF Primary Care at Lake City SW, Lake City, Florida
  - UF Primary Care at Lake City West, Lake City, Florida
  - Charles H. Croft MDPA, Melbourne, Florida
  - Daytona Heart Group, Multiple Locations, Florida
  - Southwest Florida Research Institute, Naples, Florida
  - Cardiovascular Instititute of Central Florida, Ocala, Florida
  - Ocala Research Institute Inc., Ocala, Florida
  - Orlando Health, Orlando, Florida
  - Naval Hospital Pensacola, Pensacola, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Advent Sebring, Sebring, Florida
  - James A. Haley Veterans Hospital, Tampa, Florida
  - AdventHealth Tampa - Pepin Heart Institute, Tampa, Florida
  - Interventional Cardiac Consultants, Tampa, Florida
  - BayCare Medical Group, Tampa, Florida
  - Guardian Research, Winter Park, Florida
  - Emory University, Atlanta, Georgia
  - Cardiovascular Consultants of South Georgia, LLC., Thomasville, Georgia
  - Loyola University Chicago, Chicago, Illinois
  - Medicoricium, Fairview Heights, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Midwest Cardiovascular Research and Education Foundation, Elkhart, Indiana
  - Lutheran Health Physicians, Fort Wayne, Indiana
  - Midwest Heart and Vascular Specialists, Overland Park, Kansas
  - Western Kentucky Heart And Lung, Bowling Green, Kentucky
  - The Research Group of Lexington, LLC, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Mid Michigan Health, Midland, Michigan
  - Essentia Institute of Rural Health, Duluth, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - Cardiology Associates Research. LLC, Tupelo, Mississippi
  - CHI Health Research Center, Omaha, Nebraska
  - Silver State Cardiology, Henderson, Nevada
  - The Valley Hospital, Ridgewood, New Jersey
  - Bassett Healthcare Network, Cooperstown, New York
  - NYU Langone, New York, New York
  - Weil Medical college of Cornell, New York, New York
  - Jamaica Hospital Medical Center, Richmond Hill, New York
  - Peak Clinical Trials, LLC, Apex, North Carolina
  - Pinehurst Medical Clinic, Pinehurst, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Trihealth Heart Institute, Cincinnati, Ohio
  - Heart House Research Foundation, Springfield, Ohio
  - Seton Heart Institute, Austin, Texas
  - Austin Heart, Austin, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - San Antonio Endovascular and Heart Institute, San Antonio, Texas
  - Baylor Scott and White, Temple, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Chippenham Hospital, Richmond, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - West Virginia University, Morgantown, West Virginia
- VA Caribbean Healthcare System, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ya'Qoub L, Elgendy IY, Pepine CJ. Non-obstructive Plaque and Treatment of INOCA: More to Be Learned. Curr Atheroscler Rep. 2022 Sep;24(9):681-687. doi: 10.1007/s11883-022-01044-4. Epub 2022 Jul 4. PMID 35781776
- [Derived] Handberg EM, Merz CNB, Cooper-Dehoff RM, Wei J, Conlon M, Lo MC, Boden W, Frayne SM, Villines T, Spertus JA, Weintraub W, O'Malley P, Chaitman B, Shaw LJ, Budoff M, Rogatko A, Pepine CJ. Rationale and design of the Women's Ischemia Trial to Reduce Events in Nonobstructive CAD (WARRIOR) trial. Am Heart J. 2021 Jul;237:90-103. doi: 10.1016/j.ahj.2021.03.011. Epub 2021 Mar 18. PMID 33745898

DOCUMENTS (1):
  • Informed Consent Form (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/88/NCT03417388/ICF_000.pdf